CLINICAL TRIAL: NCT04025580
Title: Systems Analyses of the Immune Response to the Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190126; 19-I-0126
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-01-31

CONDITIONS: Healthy Volunteer
Keywords: COVID-19; Systems Biology; Immunology
MeSH Terms: conditions — COVID-19 | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flucelvax, Fluvirin, or Fluzone High Dose (Experimental): Healthy Volunteer between ages 18-65 receiving Flucelvax
  Interventions: Biological: Flucelvax; Biological: Fluvirin; Biological: Fluzone High Dose

INTERVENTIONS:
Biological: Flucelvax — Seasonal influenza vaccine
Biological: Fluvirin — Seasonal influenza vaccine
Biological: Fluzone High Dose — Seasonal influenza vaccine for adults ages 65 and older

SUMMARY:
Background:

Vaccines help prevent disease by causing the body to have an immune response. Many parts of this response happen in the blood. This response happens over days and weeks after getting the vaccine. Researchers want to how the blood changes over time in response to vaccines. They want to find out why vaccines work better for some people than for others. This could help make more effective vaccines.

Objective:

To learn about how the body responds to vaccines.

Eligibility:

Healthy people ages 18 and older

Design:

Participants will be screened with a medical history, physical exam, and blood and urine tests.

Participants will have 9 visits over 6 months. All visits will include blood tests and a physical exam.

Participants will have the first visit 1 week before they get the vaccine.

Participants will get the flu vaccine at the second visit. The vaccine will be injected into the muscle of the upper arm with a needle. They will be watched for side effects for 15 minutes.

Participants will have the next 2 visits exactly 1 day and 1 week after they get the vaccine. They will have the other 5 visits about 14, 28, 70, and 100 days after they get the vaccine.

Participants will take email questionnaires about whether they had any side effects.

Participants may have optional extra study visits. These will be no more than once a month for up to 1 year after they get the vaccine. Optionally, they can also repeat the study each year through the 2023 - 2024 flu season

DETAILED DESCRIPTION:
Certain functions of the immune system are revealed only when the immune system is challenged. When a person is vaccinated, a coordinated response results: activation and interaction of distinct innate and adaptive immune cell populations and pathways, culminating in the formation of germinal centers from which antibody-producing plasma cells and memory B cells derive. By taking measurements at various time points before and after vaccination, we can build a comprehensive picture of how the immune system responds to a vaccine challenge.

The seasonal influenza vaccination provides an excellent model of coordinated immune activity involving innate and adaptive responses, as demonstrated in a past NIH study in 2009-2011; however, scientific advances and the possibility of multi-season responses in individuals warrant a new follow-up study with more comprehensive sampling. This is an open-label, prospective, exploratory study to assess the baseline and post-vaccination immune responses of healthy volunteers to an approved seasonal influenza vaccine. Subjects will undergo baseline blood collections on day -7 and on day 0 before receiving the study vaccine. After vaccination, blood will be collected on days 1, 7, 14, 28, 70, and 100. Optionally, subjects may also give blood once a month, as requested, up until 1 year after vaccination. Blood samples will be used to assess short- and long-term immunological effects of immunization. Evaluations will include vaccine antibody titers. Additional evaluations may include peripheral immune cell phenotyping, RNA sequencing (RNA-seq) of whole blood and defined peripheral blood cell subsets, and measurement of serum proteins and antibodies. Subjects may optionally provide stool samples at some visits for exploratory microbiome assessment. Additionally, subjects may optionally continue study participation annually through the 2023-24 influenza season.

The goal of this protocol is to use the collective information gathered across all healthy volunteers to understand how the immune system works as a whole.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

1. Aged 18 years and older (no upper age limit).
2. Able to provide informed consent.
3. Willing to have samples and data stored for future research.
4. Able to proficiently speak, read, and write English.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. CBC with differential, lymphocyte phenotyping with T, B, and natural killer cells (TBNK), acute care, mineral, and hepatic panels, anti-CMV immunoglobulin (Ig) G and IgM, and/or anti-Epstein-Barr virus (EBV) antibody panel values outside of the NIH Department of Laboratory Medicine normal reference ranges and deemed clinically significant by the PI at the time of screening.
2. Positive result for anti-HIV 1/2 antibody, antibody to hepatitis B surface antigen, or anti-hepatitis C virus antibody screening at the time of screening.
3. Prior receipt of a current seasonal influenza vaccine (for the season of participation).
4. History of allergy or hypersensitivity to any components of the study vaccine (e.g., egg protein, latex).
5. History of severe reactions to vaccines.
6. Use of an oral glucocorticoid within the past 30 days.
7. Receipt of a live-attenuated vaccine within the past 30 days.
8. Receipt of any experimental vaccine.
9. Receipt of any other type of vaccine (non-live and non-experimental, e.g., tetanus, diphtheria, and pertussis [TDaP]) within the past 14 days.
10. Planned vaccination before day 100 after study vaccination.
11. Current or recent use (within the past 90 days) of immunoglobulin therapy.
12. Surgery within the past 8 weeks, or planned surgery before day 100.
13. Current (within the past 30 days) treatment for active malignancy.
14. Cancer chemotherapy in the past 5 years.
15. Administration of any blood products within 90 days of the screening, or planned administration before day 100.
16. History of parasitic, amebic, fungal, or mycobacterial infections within the past 1 year with the exception of tinea pedis and onychomycosis.
17. Diabetes mellitus.
18. History of autoimmune or autoinflammatory disease.
19. History of a bleeding disorder.
20. Current use (within the past 30 days) of illicit drugs (per subject report).
21. Current use (within the past 30 days) of nicotine-containing products, including cigarettes and chewing tobacco, nicotine patches, gum, electronic cigarettes, etc.
22. Current alcohol use disorders (criteria per Diagnostic and Statistical Manual of Mental Disorders, fifth edition), within the past 30 days.
23. Serious, ongoing, uncontrolled infection within the past 30 days as per the judgement of the PI.
24. History of Guillain-Barre syndrome (GBS).
25. BMI greater than or equal to 30.
26. Known or suspected immunodeficiency within 1 year, including documented HIV infection.
27. Pregnancy or planning to become pregnant during the study period. (Women of childbearing potential must have a negative urine or serum pregnancy test at screening.)
28. Presence of conditions that, in the judgment of the PI, may put the individual at undue risk or compromise the scientific objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel D Sparks, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Result] Sparks R, Lau WW, Liu C, Han KL, Vrindten KL, Sun G, Cox M, Andrews SF, Bansal N, Failla LE, Manischewitz J, Grubbs G, King LR, Koroleva G, Leimenstoll S, Snow L; OP11 Clinical Staff; Chen J, Tang J, Mukherjee A, Sellers BA, Apps R, McDermott AB, Martins AJ, Bloch EM, Golding H, Khurana S, Tsang JS. Influenza vaccination reveals sex dimorphic imprints of prior mild COVID-19. Nature. 2023 Feb;614(7949):752-761. doi: 10.1038/s41586-022-05670-5. Epub 2023 Jan 4. PMID 36599369
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-I-0126.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Year 1 Healthy Volunteers (Pre-COVID-19); Year 2 COVID-19-recovered Individuals; Year 2 Individuals With no History of COVID-19: Healthy Volunteer between ages 18-65
  Flucelvax: Seasonal influenza vaccine
  Fluzone High Dose: Seasonal influenza vaccine for adults ages 65 and older
Period: Overall Study
Arm/Group | Year 1 Healthy Volunteers (Pre-COVID-19) | Year 2 COVID-19-recovered Individuals | Year 2 Individuals With no History of COVID-19
Started | 24 | 34 | 40
Completed | 13 | 34 | 40
Not Completed | 11 | 0 | 0
Not completed — COVID 19 restrictions at Clinical Center | 11 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Year 1 Healthy Volunteers (Pre-COVID-19) | Year 2 COVID-19-recovered Individuals | Year 2 Individuals With no History of COVID-19 | Total
Number analyzed (Participants) | 24 | 34 | 40 | 98
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 29 | 30 | 81
  >=65 years | 2 | 5 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 21 | 53
  Male | 9 | 17 | 19 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 4 | 9
  Not Hispanic or Latino | 22 | 31 | 36 | 89
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 1 | 4 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 4 | 9
  White | 12 | 30 | 28 | 70
  More than one race | 3 | 2 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 34 | 40 | 98

OUTCOME MEASURES:

1. Primary Outcome: Microneutralization Titers
Description: Change in antibody titer response to vaccination, as measured by microneutralization titers at day 0 and day 70 and its relationship with novel baseline biomarkers
Time Frame: Day 0 and Day 28 Reported in Manuscript
Population: Healthy Control and COVID-19 Recovered participants under 65 years of age for Year 2. Year 1 data not able to be generated/analyzed due to COVID-19 restrictions at the clinical center which prevented study from being completed. Year 1 samples were obtained but not analyzed and will never be analyzed.
Measure: Mean (95% Confidence Interval); unit: Log2 Fold Change
Groups:
- Year 2-Healthy Volunteers, Male, No History of COVID-19: Healthy Control Males under 65 years of age with no history of COVID-19
- Year 2-Healthy Volunteers, Female, No History of COVID-19: Healthy Control Females under 65 years of age with no history of COVID-19
- Year 2-COVID-19 Recovered Males: COVID-19 Recovered Males under 65 years of age
- Year 2-COVID-19 Recovered Females: COVID-19 Recovered Females under 65 years of age
Arm/Group | Year 2-Healthy Volunteers, Male, No History of COVID-19 | Year 2-Healthy Volunteers, Female, No History of COVID-19 | Year 2-COVID-19 Recovered Males | Year 2-COVID-19 Recovered Females
Number analyzed (Participants) | 14 | 16 | 14 | 15
Log2 Fold Change
  Fold Change for A/CNIC/1909 Strain | 0.769 [0.266 to 1.272] | 1.313 [0.517 to 2.108] | 1.716 [0.691 to 2.741] | 1.333 [0.793 to 1.874]
  Fold Change for A/HongKong/2671/2019 Strain | 1.154 [0.420 to 1.888] | 1.063 [0.464 to 1.661] | 1.501 [0.601 to 2.401] | 1.267 [0.471 to 2.063]
  Fold Change for B/Phuket/3073/2013 Strain | 0.462 [0.148 to 0.775] | 0.313 [0.057 to 0.568] | 0.929 [0.067 to 1.790] | 0.800 [0.371 to 1.229]
  Fold Change for B/Washington/02/2019 Strain | 0.308 [-0.073 to 0.689] | 0.625 [0.242 to 1.008] | 0.857 [0.045 to 1.669] | 0.800 [0.132 to 1.468]

ADVERSE EVENTS:
Time Frame: Through Day 7 post vaccination
Description: Adverse event information was collected on Day 1 and Day 7 post vaccination
Arm/Group | Flucelvax, Fluvirin, or Fluzone High Dose
All-Cause Mortality (participants affected / at risk) | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 72/98
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flucelvax, Fluvirin, or Fluzone High Dose (N=98)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (16)
Pain at Injection Site (General disorders) | 62 (62)
Headache (Nervous system disorders) | 20 (20)
Injection Site Swelling (General disorders) | 4 (4)
Injection Site Erythema (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-27): https://cdn.clinicaltrials.gov/large-docs/80/NCT04025580/Prot_SAP_000.pdf